CLINICAL TRIAL: NCT07323225
Title: Effectiveness of Combined Neural Mobilization Techniques and Capsular Stretching Exercises in Patients With Adhesive Capsulitis.
Brief Title: Neural Mobilization and Capsular Stretching in Adhesive Capsulitis
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohammad Moustafa Aldosoukki Hegazy, assisstant professor , department of health and rehabilitation sciences, college of applied medical siences, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/024/009
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; neural mobilization; capsular stretch
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: three groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neural mobilization group (Experimental): neural mobilization plus capsular stretching
  Interventions: Other: capsular stretching plus neural mobilization
- Capsular stretching group (Active Comparator): capsular stretching
  Interventions: Other: anterior, inferior and posterior capsular stretching
- Control group (Active Comparator): traditional execises
  Interventions: Other: traditional exercises

INTERVENTIONS:
Other: capsular stretching plus neural mobilization — anterior, posterior and inferior capsular stretching and neural mobilization
  Arms: Neural mobilization group
Other: anterior, inferior and posterior capsular stretching — anterior, inferior and posterior glenohumeral capsular stretching
  Arms: Capsular stretching group
Other: traditional exercises — stretching exercises for anterior GH musculture plus auto passive exercises and pendulum exercises
  Arms: Control group

SUMMARY:
Restriction of glenohumeral (GH) mobility in patients with adhesive capsulitis (AC) was known owing to capsular adhesion. There is a little evidence about the involvement of neural restriction in limiting range of motion (ROM) of the GH joint in patients with AC. Objectives: The purpose of this study is to investigate the combined effect of median nerve mobilization and capsular stretching on improving shoulder external rotation, abduction and internal rotation ROM among patients with AC. Methods Thirty patients will be randomly assigned into two equal groups : Group (A) will receive median nerve mobilization and capsular stretching while Group (B) will receive only capsular stretching (anterior, posterior and anteroinferior capsular stretching). Both groups will receive passive and self-assisted exercises. All patients in both groups will be evaluated pre and post treatment for GH external rotation, abduction and internal rotation ROM.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both gender (male &female) will be included if they would have second or third stage AC with their age between forty and seventy years
* experiencing pain, capsular adhesions, and a reduction of greater than fifty percentage in passive ROM of the GH joint (external rotation, abduction, and internal rotation compared to the sound side
* lasting for a minimum of three months. Patients with positive upper limb tension test-1 will be also included in this study

Exclusion Criteria:

* they would have stroke,Parkinson's diseases that interfere with shoulder muscles activity
* diabetes
* traumatic shoulder conditions
* glenohumeral osteoarthritis confirmed by x-ray
* previous surgery, and manipulation of the affected GH joint under general anesthesia
* Patients with passive elbow extension ROM

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 4 Weeks
  pain was assessed by VAS which has two ends. the left end indicates no pain where the right end indicates maximal pain
central sensitization | 4 weeks
  central sensitization will be assessed by the the arabic version of central sensitizatuion questionnaire. To understand CSI scores, the following severity categories have been established: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam bin Abdulaziz University, Al Kharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coppieters MW, Butler DS. Do 'sliders' slide and 'tensioners' tension? An analysis of neurodynamic techniques and considerations regarding their application. Man Ther. 2008 Jun;13(3):213-21. doi: 10.1016/j.math.2006.12.008. Epub 2007 Mar 30. PMID 17398140
- [Result] Martinez-Merinero P, Lluch E, Gallezo-Izquierdo T, Pecos-Martin D, Plaza-Manzano G, Nunez-Nagy S, Falla D. The influence of a depressed scapular alignment on upper limb neural tissue mechanosensitivity and local pressure pain sensitivity. Musculoskelet Sci Pract. 2017 Jun;29:60-65. doi: 10.1016/j.msksp.2017.03.001. Epub 2017 Mar 10. PMID 28319883